CLINICAL TRIAL: NCT03698968
Title: A Prospective Follow up Study to Assess Performance, Safety and Efficacy of the PICO 7 NPWT System for Surgically Closed Incision Sites and Skin Grafts.
Brief Title: Performance, Safety and Efficacy of PICO Device.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CT1703PC7
Record Dates: First submitted 2018-05-17; First posted 2018-10-09 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Wound Heal
Keywords: surgical complication; NPWT; negative pressure; knee arthroplasty; abdominal incision; skin graft; infection; dehisced
MeSH Terms: conditions — Infections | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Masking Description: Open
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single prospective intervention (Other)
  Interventions: Device: Negative Pressure Wound Therapy

INTERVENTIONS:
Device: Negative Pressure Wound Therapy — Single use disposable negative pressure system. The system is capable of delivering up to 80 mm Hg negative pressure to a wound or surgical incision site and managing low to moderate levels of exudate or fluid generated by the wound or incision. The therapy may be administered for up to 1 week.

SUMMARY:
The study is being conducted to evaluate the safe and effective use of the PICO 7 system in surgically closed incision sites and wounds requiring closure by skin graft or flap as part of the PMCF plan for this product, for the purpose of continuing CE (Conformité Européene) Mark approval in accordance with MEDDEV 2.12-2

DETAILED DESCRIPTION:
Although evidence exists which supports the positive effects of NPWT on take of skin grafts and flaps, there is limited evidence in relation to single-use systems such as PICO. Most previous studies have used traditional NPWT systems as part of their design. Though the technical applications of the traditional and newer single-use systems are comparable it is possible that some of the features of the latter may influence clinical outcomes. In addition to the limitations highlighted above, the cited studies have seldom assessed the ease of management and acceptability of NPWT systems. Although clinical outcomes may be considered paramount, these usability factors could also play a key role in ensuring compliance with negative pressure protocols.

Although evidence exists which supports the positive effects of NPWT on take of skin grafts and flaps, there is limited evidence in relation to single-use systems such as PICO. Most previous studies have used traditional NPWT systems as part of their design. Though the technical applications of the traditional and newer single-use systems are comparable it is possible that some of the features of the latter may influence clinical outcomes. In addition to the limitations highlighted above, the cited studies have seldom assessed the ease of management and acceptability of NPWT systems. Although clinical outcomes may be considered paramount, these usability factors could also play a key role in ensuring compliance with negative pressure protocols.

The study is being conducted to evaluate the safe and effective use of the PICO 7 system in surgically closed incision sites and wounds requiring closure by skin graft or flap as part of the PMCF plan for this product, for the purpose of continuing CE (Conformité Européene) Mark approval in accordance with MEDDEV 2.12-2.

The PICO system has recently been updated with minor modifications that make the system silent during wear. S & N also wish to collect PMCF data in the indications of knee and abdominal incisions in order to make retrospective comparisons with data previously collected for these indications.

The aim of this study is therefore to assess whether the PICO 7 system is a safe and effective therapy for surgically closed incisions, skin grafts and flaps. Effectiveness will be defined by the ability of the system to deliver negative pressure and handle exudate and by percentage of successful skin graft or flap survival at Day 14.

A summary of known and potential risks and benefits to humans of each test article can be found in the Instructions for Use of PICO 7.

ELIGIBILITY:
Inclusion Criteria:

* The subject must provide written informed consent
* Subjects eighteen (18) years of age or older.
* Willing and able to make all required study visits.
* Able to follow instructions.
* Subject is suitable to participate in the study in the opinion of the Investigator
* Subject has a suitable, closed abdominal or knee surgery incision skin flap or skin graft (STSG, meshed or non-meshed) (if there is more than one incision then the clinician should choose the one which in their opinion is most suited to PICO therapy), that fits under the absorbent dressing area of the appropriate PICO 7 dressing supplied.

Exclusion Criteria:

* Contraindications (per the PICO 7 IFU) or hypersensitivity to the use of the investigational product or their components (e.g. silicone adhesives and polyurethane films [direct contact with incision], acrylic adhesives [direct contact with skin], polyethylene fabrics and super-absorbent powders [polyacrylates]) within the dressing).
* Subjects with extremely fragile skin who require the use of SECURA non-sting barrier skin wipes and have hypersensitivity to the ingredients in the wipes
* Participation in the treatment period of another clinical trial within thirty (30) days of operative visit or during the study.
* Subjects with skin features (e.g. tattoos, skin colour, pre-existing scarring) which in the opinion of the Investigator, will interfere with the study assessments.
* Patients undergoing a procedure as part of palliative care (to be confirmed during surgery).
* Subjects with incisions or skin grafts that are actively bleeding unless haemostasis has been achieved (to be confirmed during surgery).
* Subjects with infected skin grafts or incisions at the time of surgery (except for those with perforated bowel or peritonitis).
* Subjects who have participated previously in this clinical trial
* Subjects with a history of poor compliance with medical treatment.
* Subjects with skin grafts to correct pressure ulcers where compression therapy is needed for healing (based on clinicians expertise).
* Subjects with a medical or physical condition that, in the opinion of the Investigator, would preclude safe subject participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-11-06 (Actual); Primary Completion 2019-06-18 (Actual); Study Completion 2019-06-18 (Actual)

PRIMARY OUTCOMES:
Functional clinical performance of the PICO 7 NPWT system through delivery of negative pressure | 7 Days
  Negative pressure maintenance at nominal 80 mmHg as assessed as the average of the negative pressure values recorded by the device microchip
Functional clinical performance of the PICO 7 NPWT system through wound exudate management | 7 Days
  Number of NPWT systems with no occurrence of exudate leaks as assessed through a combination of leakage alert data from device microchip and/or clinical data on any leakage observed during the dressing wearing period resulting or not, in an unplanned dressing change
Composite Clinical Success | 7 Days
  Composite Clinical Success (CCS) defined as a binary variable (1/0) (1 if both of the following are true and 0 if at least one of the two is false):
  A. Nominal pressure is in the interval 80mmHg ± 7mmHg
  B. No leakage

SECONDARY OUTCOMES:
Number of participants with incidence of Surgical Site Infection (SSI) - Superficial, deep. [CDC criteria] | 30 Days
  For incidence of SSI and incidence of SSC binary variables indicating presence of/absence of will be defined and the frequencies together with percentages reported/identified outcomes will be reported. Logistic models will be fitted and associated factors adjusted for if there is adequate data
Number of participants with incidence of Surgical Site Complications (SSC) - dehiscence (superficial/deep etc.), seroma, necrosis, hematoma, suture abscess | 30 Days
  For incidence of SSI and incidence of SSC binary variables indicating presence of/absence of will be defined and the frequencies together with percentages reported/identified outcomes will be reported. Logistic models will be fitted and associated factors adjusted for if there is adequate data
Percentage of successful skin graft take or flap survival at Days 7, 14 and 30 | 30 Days
  Assessed by clinician visual assessment
Visual inspection of peri-wound skin condition | 30 Days
  Visual inspection assessment (e.g., healthy, fragile, inflamed, erythema, bruising, eczematous, dry/flaky, macerated) at 7, 14 and 30 days
Visual Analog Scale (VAS) - pain | 30 Days
  Level of subject pain during wear of the PICO 7 system, at dressing removal and at application assessed by VAS scale (pain intensity as none, mild, moderate, or severe) following 7 day therapy
Dressing wear time in days | 30 Days
  Assessed through a combination of data from device microchip and CRF recorded data of any unplanned dressing change

CONTACTS AND LOCATIONS:
Overall Officials: Rachael Winter, Study Director — T.J. Smith & Nephew, LTD; Sudheer Karlakki, Principal Investigator — Robert Jones & Agnes Hunt Orthopaedic Hospital
Locations (11):
- Ospedale Regionale di Lugano; Sede Ospedale Italiano, Lugano, Switzerland
- United Kingdom (10):
  - Mid Essex Hospital Services, Chelmsford, Essex
  - The Robert Jones & Agnes Hunt Orthopaedic Hospital NHS Foundation, Oswestry, Shropshire
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Queen Victoria Hospital, East Grinstead
  - Manchester University NHS Foundation Trust, Manchester
  - Queen Elizabeth the Queen Mother Hospital, Margate
  - North Tyneside General Hospital, North Shields
  - Norfolk & Norwich University Hospital, Norwich
  - Peterborough City Hospital, North West Anglia NHS Foundation Trust, Peterborough
  - Mid-Yorkshire NHS Trust, Wakefield